CLINICAL TRIAL: NCT05771909
Title: Effect of App-driven Deep Breathing (NEURODIGITX) on Anxiety Levels and Quality of Life in Caregivers: a Randomized Controlled Trial
Brief Title: Effect of App-driven Deep Breathing (NEURODIGITX) on Anxiety Levels and Quality of Life in Caregivers
Acronym: DIAL_X
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: medical device not available
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DIAL_X
Record Dates: First submitted 2023-02-24; First posted 2023-03-16 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Disorders; Hospital Workers; Deep Breath
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NeurodigitX (Experimental): After randomization, the "NeurodigitX Group" receiving this program will follow the recommendations for a period of three months (2 sessions of 2 minutes per day).
  At this visit and at the 1/2/3 and 6 month visits, staff will complete the following scales and questionnaires (15 minutes in length): Visual Anxiety Analog Scale (VAS), Spielberger Anxiety Scale - State (STAI form Y-A) and SF-12 Quality of Life Questionnaire.
  All participants will be called in at 3 months for a visit to measure HRV via the app.
  Interventions: Other: NeurodigitX
- Control (Other): After randomization, the "Control Group" does not receive the NeurodigitX application.
  At this visit and at the 1/2/3 and 6 month visits, staff will complete the following scales and questionnaires (15 minutes in length): Visual Anxiety Analog Scale (VAS), Spielberger Anxiety Scale - State (STAI form Y-A) and SF-12 Quality of Life Questionnaire.
  All participants will be called in at 3 months for a visit to measure HRV via the app.
  Interventions: Other: Control

INTERVENTIONS:
Other: NeurodigitX — The "NeurodigitX Group" receiving this program will follow the recommendations for a period of three months (2 sessions of 2 minutes per day).
  Arms: NeurodigitX
Other: Control — The "Control Group" does not receive the NeurodigitX application.
  Arms: Control

SUMMARY:
The occurrence of the COVID-19 pandemic is associated with an increase in psychiatric illnesses (depression, anxiety) in the general population due to the infectious and vital risk involved, changes in social structure, particularly in the family environment, episodes of confinement, and even professional instability. These international phenomena have also been observed in France.

In addition to the constraints of the general population, health care workers have been, and continue to be, subject to other forms of constraints, linked to their professional activity. Indeed, the risk of viral exposure is for them major, the confrontation with the deaths of patients because of their fragility or the weakness of the care structures, are more violent in connection with their immediate reality. In addition, the workload due to health imperatives has also led to physical and psychological exhaustion of the health care teams. In addition to the international evidence, the existence and severity of the psychological consequences for health care workers have recently been documented at the local level in a survey conducted among the staff of the Groupe hospitalier Paris Saint-Joseph (GhPSJ). In this study of more than 780 people, nearly half of whom were in charge of patients infected with SARS-CoV2, 62% reported increased anxiety since the beginning of the epidemic, 41% had symptoms of anxiety, 21% had symptoms of depression and 14% had signs of post-traumatic stress. Approximately 25% of the total population had chosen to make regular use of the "bulle" (a decompression and care platform made available to staff since the first wave within the establishment) with the aim of reducing the anxiety generated by the situation and particularly by their professional activity. Given the importance of anxiety symptoms detected in healthcare professionals during the COVID-19 pandemic, the use of a simple, brief technique, requiring neither trained personnel nor expensive or difficult-to-access devices, aimed at reducing anxious stress could be of significant benefit to the population, especially to caregivers.

The objective of this study is to measure the effect of deep breathing on the anxiety of health professionals in the aftermath of the COVID-19 pandemic, and its effect on their quality of life. In order to measure the quality of the sessions, the breathing movements will be performed using a calibrated program and their immediate effectiveness will be evaluated by the variation of the heart rate, visible just after the program by the user.

The NeurodigitX® system offers to control interactive 3D games on a smartphone application through breath via a sensor connected to the phone by Bluetooth. This tool also allows to measure by plethysmography the heart rate variability in a simple and non-invasive way.

This system has been created as a preventive health solution by allowing everyone to measure, compare and share the activity of their Autonomic Nervous System (ANS) to better predict, understand, prevent and treat certain chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthcareworkers whose age ≥ 18 years,
* Healthcareworkers working in the Emergency Department, Intensive Care Unit and/or visiting the Bulle at least once a week (frequency assessed by Delphi method) at Hôpital Paris Saint-Joseph, healthcareworkers visiting the Bulle at Hôpital Marie-Lannelongue at least once a week and healthcareworkers working at Hôpital Sainte-Marie or Hôpital Léopold Bellan
* French speaking staff
* Staff affiliated to the social security system or, failing that, to another health insurance system
* Staff who have given their free, informed and written consent

Exclusion Criteria:

* Current participation in another interventional study regarding post-traumatic stress or anxiety
* Regular practice in the last year of deep breathing techniques in the context of anxiety management (meditation, cardiac coherence, etc.)
* Use of medications that slow down the heart rate: antiarrhythmics, calcium channel blockers, beta-blockers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-11-29 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of a 3-month program of regular deep breathing practice on anxiety | Month 3
  This outcome corresponds to the comparison of the evolution of anxiety scores between the 2 groups NeuroDigitX and Control, by Spielberger's State-Trait Anxiety Inventory. Each response to a STAI item is scored from 1 to 4, with 1 indicating the lowest degree of anxiety and 4 the highest. For the AE and AT scales, there are 10 and 9 items respectively. To obtain the AE score, the scores obtained on the 20 items corresponding to AE (items 1 to 20) are added together.

SECONDARY OUTCOMES:
Effect of the program on quality of life at 3 month | Month 3
  This outcome corresponds to the comparison of changes in quality of life scores. The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  The SF-12 is a shortened version of it's predecessor, the SF-36, which itself evolved from the Medical Outcomes Study. The SF-12 was created to reduce the burden of response.
Effect of the program on quality of life at 6 month | Month 6
  This outcome corresponds to the comparison of changes in quality of life scores.The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  The SF-12 is a shortened version of it's predecessor, the SF-36, which itself evolved from the Medical Outcomes Study. The SF-12 was created to reduce the burden of response.
Effect of the program on the evolution of heart rate variability at 3 month | Month 3
  This outcome corresponds to the comparison of changes in heart rate variability measurements between the 2 groups at 3 months.
Effect of the program by profession and department (emergency, intensive care, other department) | Day 1
  This outcome corresponds to the comparison of measures of anxiety according to the occupation and service of the volunteers.
Effect of the program by profession and department (emergency, intensive care, other department) | Month 6
  This outcome corresponds to the comparison of measures of anxiety according to the occupation and service of the volunteers. Spielberger's State-Trait Anxiety Inventory: Each response to a STAI item is scored from 1 to 4, with 1 indicating the lowest degree of anxiety and 4 the highest. For the AE and AT scales, there are 10 and 9 items respectively. To obtain the AE score, the scores obtained on the 20 items corresponding to AE (items 1 to 20) are added together.

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite D'USSEL, MD, Study Director — Fondation Hôpital Saint-Joseph
Locations (4):
- France (4):
  - Hôpital Marie Lannelongue, Le Plessis-Robinson
  - Hôpital Léopold BELLAN, Paris
  - Hôpital Paris Saint-Joseph, Paris
  - Hôpital Sainte-Marie, Paris

REFERENCES:
- [Background] Casagrande M, Favieri F, Tambelli R, Forte G. The enemy who sealed the world: effects quarantine due to the COVID-19 on sleep quality, anxiety, and psychological distress in the Italian population. Sleep Med. 2020 Nov;75:12-20. doi: 10.1016/j.sleep.2020.05.011. Epub 2020 May 12. PMID 32853913
- [Background] Choi EPH, Hui BPH, Wan EYF. Depression and Anxiety in Hong Kong during COVID-19. Int J Environ Res Public Health. 2020 May 25;17(10):3740. doi: 10.3390/ijerph17103740. PMID 32466251
- [Background] Dutheil F, Mondillon L, Navel V. PTSD as the second tsunami of the SARS-Cov-2 pandemic. Psychol Med. 2021 Jul;51(10):1773-1774. doi: 10.1017/S0033291720001336. Epub 2020 Apr 24. PMID 32326997
- [Background] Ozamiz-Etxebarria N, Dosil-Santamaria M, Picaza-Gorrochategui M, Idoiaga-Mondragon N. Stress, anxiety, and depression levels in the initial stage of the COVID-19 outbreak in a population sample in the northern Spain. Cad Saude Publica. 2020 Apr 30;36(4):e00054020. doi: 10.1590/0102-311X00054020. eCollection 2020. English, Spanish. PMID 32374806
- [Background] Serafini G, Parmigiani B, Amerio A, Aguglia A, Sher L, Amore M. The psychological impact of COVID-19 on the mental health in the general population. QJM. 2020 Jun 22;113(8):531-7. doi: 10.1093/qjmed/hcaa201. Online ahead of print. PMID 32569360
- [Background] d'Ussel M, Fels A, Durand X, Lemogne C, Chatellier G, Castreau N, Adam F. Factors associated with psychological symptoms in hospital workers of a French hospital during the COVID-19 pandemic: Lessons from the first wave. PLoS One. 2022 Apr 28;17(4):e0267032. doi: 10.1371/journal.pone.0267032. eCollection 2022. PMID 35482772
- [Background] d'Ussel M, Adam F, Fels A, Chatellier G, Philippart F. Characteristics of Hospital Workers Using a Wellbeing Center Implemented During the COVID-19 Pandemic to Prevent the Emotional Impacts of the Crisis. Front Public Health. 2022 Jul 4;10:913126. doi: 10.3389/fpubh.2022.913126. eCollection 2022. PMID 35859769
- [Background] Lefevre H, Stheneur C, Cardin C, Fourcade L, Fourmaux C, Tordjman E, Touati M, Voisard F, Minassian S, Chaste P, Moro MR, Lachal J. The Bulle: Support and Prevention of Psychological Decompensation of Health Care Workers During the Trauma of the COVID-19 Epidemic. J Pain Symptom Manage. 2021 Feb;61(2):416-422. doi: 10.1016/j.jpainsymman.2020.09.023. Epub 2020 Sep 19. PMID 32961219